CLINICAL TRIAL: NCT00120133
Title: Use of Atorvastatin (Lipitor) to Prevent Bone Pain Following Infusion of Pamidronate or Zoledronic Acid
Brief Title: Atorvastatin (Lipitor) to Prevent Bone Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: #04 10-119
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2005-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bisphosphonates; Atorvastatin
MeSH Terms: conditions — Osteoporosis | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
In the proposed randomized double blind cross-over placebo controlled study, the researchers intend to investigate if Atorvastatin (FDA approved statin for children) can be used to alleviate the symptom of bone pain (acute phase reaction) that is commonly associated with initial doses of pamidronate or zoledronic acid, and also the mechanism that underlies this proposed beneficial effect of Atorvastatin. The primary outcome studied will be alleviation of bone pain by Atorvastatin compared to placebo by visual analogue pain scale in children treated with pamidronate or zoledronic acid. The secondary outcome investigated will be changes in blood count and γδT cell count, C-reactive protein (CRP) and cytokine levels of interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and gamma interferon (γ-IFN) following treatment with Atorvastatin compared to placebo.

DETAILED DESCRIPTION:
The proposed study is a double blind cross-over placebo controlled randomized clinical study that would be conducted in the Metabolic Bone Clinic of The Children's Mercy Hospital. This is a pilot study and a more comprehensive study will be designed only if the results from this pilot study are significant. In our proposed double blind cross-over placebo controlled pilot study we will have a total of 12 children who will receive either placebo or Atorvastatin in a randomized cross-over design. The pilot study with a sample of 12 in a cross-over trial will provide reasonably stable estimates even though it is unlikely to provide statistical significance on its own but will help plan further large scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Children with various metabolic bone diseases and osteoporosis who are to initiate treatment with either pamidronate and/or zoledronic acid.
* They should be 6 to 25 years old, able to understand the study, swallow pills and competent to complete the visual analogue pain scale.

Exclusion Criteria:

* Children less than 6 years old or incompetent to complete the visual analogue pain scale.
* Children with seizure disorder associated or triggered by fever.
* Children known to have hypersensitivity reaction to statins, active liver disease or persistent elevated serum transaminases or CPK.
* Children on erythromycin, cyclosporine, fibric acid, azole antifungals, cimetidine and spironolactone will be excluded.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2004-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Alleviation of bone pain by Atorvastatin compared to placebo by visual analogue pain scale.

SECONDARY OUTCOMES:
Changes in blood count and γδT cell count, CRP and cytokine levels of interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α) and gamma interferon (γ-IFN) following treatment with Atorvastatin compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Tarak Srivastava, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Srivastava T, Haney CJ, Alon US. Atorvastatin may have no effect on acute phase reaction in children after intravenous bisphosphonate infusion. J Bone Miner Res. 2009 Feb;24(2):334-7. doi: 10.1359/jbmr.081016. PMID 18847329